CLINICAL TRIAL: NCT06611696
Title: Avacopan With Short-term Reduced-dose Glucocorticoids vs Reduced-dose Glucocorticoids Added to Rituximab on Remission Induction in ANCA-associated Vasculitis
Brief Title: Avacopan vs Reduced-dose Glucocorticoids in ANCA-associated Vasculitis
Acronym: ARRIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chiba University (Other)
Collaborators: Kissei Pharmaceutical Co., Ltd. (Industry); International University of Health and Welfare (Other)
Responsible Party: Principal Investigator, Shunsuke Furuta, Associate Professor, Department of Allergy and Clinical Immunology, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRB0097-24
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-11

CONDITIONS: ANCA Associated Vasculitis (AAV)
Keywords: microscopic polyangiitis; granulomatosis with polyangiitis; avacopan; ANCA-associated vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Granulomatosis with Polyangiitis | interventions — avacopan; Prednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucocorticoid group (Active Comparator): Prednisolone will be commenced with dose of 0.5mg/kg/day and will be tapered and off within 5 months. If a patient fails to achieve BVAS=0 or normalization of CRP levels or normalization of ANCA levels, an investigator can keep 5mg/day of prednisolone and postpone the procedure of stopping prednisolone. Patients will also receive rituximab (375mg/m2/w x4).
  During remission maintenance phase (6-24 months),, patients will receive rituximab (500mg/body) every 6 months as remission maintenance therapy.
  In the case of inadequate response to the combination therapy of prednisolone and rituximab, additional administration of prednisolone 20mg/day (less than 2 weeks) can be allowed as the rescue therapy.
  During remission maintenance phase, in the case of minor relapse, additional administration of prednisolone 20mg/day (less than 2 weeks) can be allowed as the rescue therapy. Minor relapse is defined as relapse with no major BVAS item.
  Interventions: Drug: Prednisolone and rituximab
- Avacopan group (Experimental): Prednisolone will be commenced with dose of 0.5mg/kg/day and will be tapered and off within 1 months. Patients will also receive avacopan (60mg/day) and rituximab (375mg/m2/w x4).
  During remission maintenance phase (6-24 months), patients will receive avacopan (60mg/day) as remission maintenance therapy until the trial end.
  In the case of inadequate response to the combination therapy of avacopan, prednisolone and rituximab, additional administration of prednisolone 20mg/day (less than 2 weeks) can be allowed as the rescue therapy.
  During remission maintenance phase, in the case of minor relapse, additional administration of prednisolone 20mg/day (less than 2 weeks) can be allowed as the rescue therapy. Minor relapse is defined as relapse with no major BVAS item.
  Interventions: Drug: Avacopan, prednisolone and rituximab

INTERVENTIONS:
Drug: Avacopan, prednisolone and rituximab — Patients in the avacoapn group will be treated with avacoapn, short-term reduced-dose prednisolone and rituximab.
  Arms: Avacopan group
Drug: Prednisolone and rituximab — Patients in the glucocorticoid arm will be treated with reduced-dose prednisolone and rituximab.
  Arms: Glucocorticoid group

SUMMARY:
The goal of this clinical trial is to learn if avacopan in combination with short-term (4 weeks) reduced-dose glucocorticoid and rituximab works to treat patients with newly-onset ANCA-associated vasculitis. It will also learn about the long-term safety of avacopan. The main questions it aims to answer are:

Is avacopan in combination with short-term reduced-dose glucocorticoid and rituximab as effective as the combination of 20 week reduced-dose glucocorticoid and rituximab in the proportion of the patients achieving remission? Does avacopan lower the relapse rate compared to the 6 monthly rituximab maintenance therapy? What medical problems do participants have when taking long-term avacopan?

Participants will:

Be treated with avacopan in combination with short-term (until 4 weeks) reduced-dose glucocorticoid and rituximab (at 0 week) or reduced-dose glucocorticoid (until 20 weeks) and rituximab (at 0, 26, 52 and 78 weeks).

Be assessed at 0, 4, 8, 16, 26, 52, 78 and 104 weeks regarding disease status (remission/relapse), disease activity by Birmingham Vasculitis Activity Score ver3, disease damage by Vasculitis Damage Index and adverse events.

The primary endpoint is remission rates at 26 weeks.

DETAILED DESCRIPTION:
Anti-neutrophil cytoplasm antibody (ANCA)-associated vasculitis is characterized by a small to medium-size vasculitis and the presence of ANCA. ANCA-associated vasculitis includes microscopic polyangiitis, granulomatosis with polyangiitis and eosinophilic granulomatosis with polyangiitis. ANCA-associated vasculitis can be a life-threatening disease and the mortality is 80% at 1 year in untreated patients. In 2010s, standard therapies for remission induction of ANCA-associated vasculitis were the combination of high-dose glucocorticoids and either cyclophosphamide or rituximab. Although those therapies have high remission rates of 80-90%, mortality at 5 years is still high at 10-20% mainly due to treatments-related adverse events.

In the LoVAS trial (2021, JAMA), the combination of reduced-dose glucocorticoid and rituximab showed non-inferiority to high-dose glucocorticoid and rituximab in remission rates at 6 months. In addition, adverse events were dramatically less in the reduced-dose group than in the high-dose group.

In the ADVOCATE trial (2021, NEJM), the combination of avacopan, newly developed complement C5a inhibitor, and rituximab or cyclophosphamide showed non-inferiority to high-dose glucocorticoid and rituximab or cyclophosphamide in remission rates at 6 months. The avacopan group was allowed to use glucocorticoid within 1 month from the trial entry, and over 80% of patients used glucocorticoid indeed. Regarding adverse events, they were less in the avacopan group than in the glucocorticoid group.

Although both the reduced-dose glucocorticoid regimen in the LoVAS trial and the avacopan regimen in the ADVOCATE trial are effective and safe for patients with ANCA-associated vasculitis, there is no trial directly comparing both regimens at the moment. Thus, in this multicenter, open-label, randomized, non-ineriority, phase 4 trial, the investigators aim to investigate if the combination of avacoapn, short-term (4 weeks) reduced-dose glucocorticoid and rituximab is non-inferior to the combination of reduced-dose glucocorticoid (20 weeks) and rituximab. The investigators also compare safety profiles and disease relapse between the two groups. A total of 160 patients with new-onset ANCA-associated vasculitis (microscopic polyangiitis and granulomatosis with polyangiitis) will be recruited and randomized to the two treatments groups. The primary end point is remission rate at 26 weeks, and the patients will be followed until 104 weeks for assessing disease relapse and long-term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent by a patient or a surrogate decision maker
2. Age=>18 years
3. New clinical diagnosis of ANCA-associated vasculitis (granulomatosis with polyangiitis, microscopic polyangiitis) consistent with the 2012 Chapel Hill consensus definitions and 2022 EULAR/ACR classification criteria
4. Positive test by ELISA, CLEIA or FEIA for proteinase 3-ANCA or myeloperoxidase-ANCA

Exclusion Criteria:

1. Prior treatment for ANCA-associated vasculitis before trial entry
2. ANCA-associated vasculitis related glomerulonephritis (eGFR less than 15ml/min) or alveolar hemorrhage (oxygen inhalation more than 2L/min)
3. Presence of another multisystem autoimmune disease
4. Known infection with HIV; a past or current history of hepatitis B virus or hepatitis C virus infection
5. Desire to bear children, pregnancy or lactating
6. History of malignancy within the past 5 years or any evidence of persistent malignancy
7. Ongoing or recent (last 1 year) evidence of active tuberculosis
8. History of severe allergy or anaphylaxis to monoclonal antibody therapy
9. Any concomitant condition anticipated to likely require oral systemic glucocorticoids, immunosuppressants, biologics, plasma exchange or IVIg
10. Any biological B cell depleting agent (such as rituximab or belimumab)-use within the past 6 months
11. Past history of medication of avacopan
12. Patients can not take avacopan and prednisolone orally
13. Other conditions, in the investigator's opinion, inappropriate for the trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportions of patients achieving remission | 26 weeks
  Remission is defined as BVAS (Birmingham vasculitis activity score)=0 and less than 5mg/day of prednisolone.

SECONDARY OUTCOMES:
Sustained remission without taking prednisolone at 104 weeks | 104 weeks
  Remission is defined as BVAS (Birmingham vasculitis activity score)=0 and less than 5mg/day of prednisolone.
Survival, relapse and end-stage renal disease | 26 and 104 weeks
  Assessed by Kaplan-Meier curves.
Accumulative dose of glucocorticoids | 26 and 104 weeks
  Accumulative dose of glucocorticoids during the study period
Birmingham Vasculitis Activity Score (BVAS) version 3 | 26 and 104 weeks
  BVAS is a scoring system for assessing the disease activity of vasculitis.
Vasculitis Damage Index (VDI) | 104 weeks
  VDI is a scoring system for assessing irreversible disease damage due to vasculitis.
Short-Form 36 (SF-36) | 26 and 104 weeks
  SF-36 is a scoring system for assessing patient QOL.
Serious adverse event (SAE) | 26 and 104 weeks
  Event numbers and proportions of patients with one or more SAEs.
Proportions of the patients with new onset diabetes mellitus | 26 and 104 weeks
  Diabetes mellitus requiring drug treatments
Proportions of the patients with new onset hypertension | 26 and 104 weeks
  Hypertension requiring drug treatments
Proportions of the patients with new onset hyperlipidemia | 26 and 104 weeks
  Hyperlipidemia requiring drug treatments
Proportion of the patients with new onset bone fracture, bone density | 104 weeks
  Bone density is assessed at lumber spines.
Number of infections, proportions of the patients with infection | 26 and 104 weeks
  Infections requiring drug treatments
Number of serious infections, proportions of the patients with serious infection | 26 and 104 weeks
  Serious infections are serious events among infections requiring drug treatments.
Proportions of the patients with liver dysfunction | 26 and 104 weeks
  Liver dysfunction >= grade 3 liver dysfunction (CTCAE)
Proportions of the patients with new onset malignancies | 26 and 104 weeks
  Malignancies diagnosed after the trial entry
Proportions of patients achieving remission without the rescue therapy | 26 weeks
  Remission is defined as BVAS (Birmingham vasculitis activity score)=0 and less than 5mg/day of prednisolone.
Sustained remission without taking prednisolone at 104 weeks and the rescue therapy during the trial period | 104 weeks
  Remission is defined as BVAS (Birmingham vasculitis activity score)=0 and less than 5mg/day of prednisolone.
Proportions of patients treated with the rescue therapy | 26 and 104 weeks
  Details of the rescue therapy are written in the section of "Arms and Interventions".

CONTACTS AND LOCATIONS:
Overall Officials: Masayoshi Harigai, MD, PhD, Principal Investigator — International University of Health and Welfare
Locations (22):
- Japan (22):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - Chiba Aoba Municipal Hospital, Chiba, Chiba
  - Chiba University, Chiba, Chiba
  - Chiba Rosai Hospital, Ichihara, Chiba
  - Kameda Medical Centre, Kamogawa, Chiba
  - International University of Health and Welfare, Narita, Chiba
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - Gunma University, Maebashi, Gunma
  - Kagawa University, Hiragi, Kagawa-ken
  - St.Marianna University School of Medicine, Kawasaki, Kanagawa
  - Tohoku Univerisity, Sendai, Miyagi
  - Nagasaki University, Nagasaki, Nagasaki
  - Okayama University, Okayama, Okayama-ken
  - Kitano Hospital, Osaka, Osaka
  - Saitama Medical University, Kawagoe, Saitama
  - Dokkyo Medical University, Mibu, Tochigi
  - Juntendo Univeristy, Bunkyoku, Tokyo
  - Kyorin University, Mitaka, Tokyo
  - Toho University, Ōta-ku, Tokyo
  - Teikyo University, tabashi City, Tokyo
  - Yamanashi University, Chuo-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP
Time Frame: After publishing the report regarding all the pre-defined trial data.
Access Criteria: Data requests should be sent to Dr Shunsuke Furuta at shfuruta@chiba-u.jp or Dr Masayoshi Harigai at mharigai@iuhw.ac.jp. The requests should be assessed and permitted according to the individual purposes of the requests.
URL: https://www.m.chiba-u.jp/dept/allergy-clin-immunol/researcher/clinical/

REFERENCES:
- [Background] Exley AR, Bacon PA, Luqmani RA, Kitas GD, Gordon C, Savage CO, Adu D. Development and initial validation of the Vasculitis Damage Index for the standardized clinical assessment of damage in the systemic vasculitides. Arthritis Rheum. 1997 Feb;40(2):371-80. doi: 10.1002/art.1780400222. PMID 9041949
- [Background] Mukhtyar C, Lee R, Brown D, Carruthers D, Dasgupta B, Dubey S, Flossmann O, Hall C, Hollywood J, Jayne D, Jones R, Lanyon P, Muir A, Scott D, Young L, Luqmani RA. Modification and validation of the Birmingham Vasculitis Activity Score (version 3). Ann Rheum Dis. 2009 Dec;68(12):1827-32. doi: 10.1136/ard.2008.101279. Epub 2008 Dec 3. PMID 19054820
- [Background] Suppiah R, Robson JC, Grayson PC, Ponte C, Craven A, Khalid S, Judge A, Hutchings A, Merkel PA, Luqmani RA, Watts RA; DCVAS INVESTIGATORS. 2022 American College of Rheumatology/European Alliance of Associations for Rheumatology classification criteria for microscopic polyangiitis. Ann Rheum Dis. 2022 Mar;81(3):321-326. doi: 10.1136/annrheumdis-2021-221796. Epub 2022 Feb 2. PMID 35110332
- [Background] Robson JC, Grayson PC, Ponte C, Suppiah R, Craven A, Judge A, Khalid S, Hutchings A, Watts RA, Merkel PA, Luqmani RA; DCVAS Investigators. 2022 American College of Rheumatology/European Alliance of Associations for Rheumatology classification criteria for granulomatosis with polyangiitis. Ann Rheum Dis. 2022 Mar;81(3):315-320. doi: 10.1136/annrheumdis-2021-221795. Epub 2022 Feb 2. PMID 35110333
- [Background] Hellmich B, Sanchez-Alamo B, Schirmer JH, Berti A, Blockmans D, Cid MC, Holle JU, Hollinger N, Karadag O, Kronbichler A, Little MA, Luqmani RA, Mahr A, Merkel PA, Mohammad AJ, Monti S, Mukhtyar CB, Musial J, Price-Kuehne F, Segelmark M, Teng YKO, Terrier B, Tomasson G, Vaglio A, Vassilopoulos D, Verhoeven P, Jayne D. EULAR recommendations for the management of ANCA-associated vasculitis: 2022 update. Ann Rheum Dis. 2024 Jan 2;83(1):30-47. doi: 10.1136/ard-2022-223764. PMID 36927642
- [Background] Furuta S, Nakagomi D, Kobayashi Y, Hiraguri M, Sugiyama T, Amano K, Umibe T, Kono H, Kurasawa K, Kita Y, Matsumura R, Kaneko Y, Ninagawa K, Hiromura K, Kagami SI, Inaba Y, Hanaoka H, Ikeda K, Nakajima H; LoVAS Collaborators. Effect of Reduced-Dose vs High-Dose Glucocorticoids Added to Rituximab on Remission Induction in ANCA-Associated Vasculitis: A Randomized Clinical Trial. JAMA. 2021 Jun 1;325(21):2178-2187. doi: 10.1001/jama.2021.6615. PMID 34061144
- [Background] Jayne DRW, Merkel PA, Schall TJ, Bekker P; ADVOCATE Study Group. Avacopan for the Treatment of ANCA-Associated Vasculitis. N Engl J Med. 2021 Feb 18;384(7):599-609. doi: 10.1056/NEJMoa2023386. PMID 33596356
- [Background] Jennette JC, Falk RJ, Bacon PA, Basu N, Cid MC, Ferrario F, Flores-Suarez LF, Gross WL, Guillevin L, Hagen EC, Hoffman GS, Jayne DR, Kallenberg CG, Lamprecht P, Langford CA, Luqmani RA, Mahr AD, Matteson EL, Merkel PA, Ozen S, Pusey CD, Rasmussen N, Rees AJ, Scott DG, Specks U, Stone JH, Takahashi K, Watts RA. 2012 revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides. Arthritis Rheum. 2013 Jan;65(1):1-11. doi: 10.1002/art.37715. No abstract available. PMID 23045170
- See also: English version of the protocol is now preparing and will be shown in the above website. — https://www.m.chiba-u.jp/dept/allergy-clin-immunol/researcher/clinical/
- Available data/document: Study Protocol — https://www.m.chiba-u.jp/dept/allergy-clin-immunol/researcher/clinical/ — Regarding deidentified patient data, please request to Dr Shunsuke Furuta at shfuruta@chiba-u.jp or Dr Masayoshi Harigai at mharigai@iuhw.ac.jp after publishing pre-defined trial results.